CLINICAL TRIAL: NCT02641197
Title: Vascular Reactivity Assessment by AngioDefender -- A Repeatability and Reproducibility Study
Brief Title: Vascular Reactivity Assessment by the AngioDefender Device -- A Precision Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Everist Genomics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A-1501
Record Dates: First submitted 2015-12-16; First posted 2015-12-29 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Cardiovascular Diseases
Keywords: flow-mediated dilation; AngioDefender; device precision; repeatability; reproducibility; cardiovascular diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AngioDefender (Experimental): The AngioDefender device uses a novel, proprietary software algorithm to analyze pulse wave amplitude data collected before and after brachial artery occlusion by a standard upper arm pneumatic blood pressure cuff. The procedure is non-invasive and does not employ ultrasound.
  Interventions: Device: AngioDefender

INTERVENTIONS:
Device: AngioDefender — Repeatability will be assessed by repeat AngioDefender (AD) testing of the same subject 1 hour apart, using the same AD device and operator.
  Reproducibility will be assessed by comparing FMD scores obtained for the same subject, but using different AD devices and operators.

SUMMARY:
The objective of this study is to define the repeatability and reproducibility of quantifying flow-mediated dilation (FMD) of the brachial artery (BA) using the AngioDefender (AD) methodology.

Repeatability will be assessed by repeat AD testing of the same subject 1 hour apart, using the same AD device and operator.

Reproducibility will be assessed by comparing FMD scores obtained for the same subject, but using different AD devices and operators.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ≥18 years old
2. Eastern Cooperative Oncology Group/Zubrod score performance status of 0, 1, or 2, determined within 7 days prior to FMD testing on Study Day 1 (Visit 1)
3. Written informed consent understood and signed; understanding of study procedures and ability to comply with them for the length of the study

Exclusion Criteria:

1. Body mass index (BMI) >50 kg/m2
2. Mid-upper arm circumference of arm selected for FMD testing <17 cm or >42 cm
3. Sinus arrhythmia, atrial fibrillation, atrial flutter, multifocal atrial tachycardia, frequent (>1 per 10-sec strip) premature atrial or ventricular contractions (isolated, non-isolated, or alternating), documented by 12-lead ECG with rhythm strip at the time of subject screening.
4. Clinical signs and/or symptoms of active viral or bacterial infections
5. Resting muscle tremor or inability to remain still for the duration of the testing period
6. Systolic blood pressure (SBP) at rest of >170 mmHg or diastolic blood pressure (DBP) at rest of ≥110 mmHg.
7. Diabetic subjects - Type I or II
8. Previous intolerable adverse reaction(s) to vascular testing using an upper extremity occlusive pneumatic cuff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-06 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline %flow-mediation dilation (%FMD) at 1 hour | Daily x 4 consecutive days
  Repeat AD testing of the same subject 1 hour apart on 4 consecutive days (operators and/or AD devices change each day)

SECONDARY OUTCOMES:
Reproducibility of multiple %FMD determinations by AngioDefender | Daily x 4 consecutive days
  Repeat AD testing of the same subject over 4 consecutive days using different operators and/or AD devices each day
Incidence of emergent adverse device effects (ADEs) according to CTCAE v4.03 | 4 consecutive days (maximum 5 days)
  Spontaneous ADEs reported by the subject and inquiry into emergence of expected/unexpected ADEs

CONTACTS AND LOCATIONS:
Overall Officials: Peter F Lenehan, MD PhD, Study Director — Everist Genomics, Inc
Locations (2):
- Canada (2):
  - University of Western Ontario, London, Ontario
  - Hotel-Dieu Grace Healthcare, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No